CLINICAL TRIAL: NCT00188604
Title: A Randomized Phase II Placebo-controlled Double Blind Study of Using Selenium in the Treatment of Secondary Lymphedema in Breast Cancer Patients
Brief Title: The Use of Selenium to Treat Secondary Lymphedema - Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UHN REB 03-0741-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Breast Neoplasms; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Sodium Selenite

INTERVENTIONS:
Drug: sodium selenite

SUMMARY:
The primary objective of this study to assess the effectiveness of selenium compared to placebo in reducing the lymphedema in-patients with breast cancer. Secondary objectives are to assess the impact of selenium on patient's quality of life and to assess the incidence of adverse effects of selenium therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically documented lymphedema of upper limb secondary to breast cancer management (surgery - axillary nodal dissection, and radiotherapy)
* patients who have had other modalities of management can be included, e.g. physical therapy, pharmacological therapy
* ECOG performance 0-2
* informed consent

Exclusion Criteria:

* active cellulitis/skin infection of the limb
* venous thrombosis of the upper limbs
* active malignancy
* any other medical condition or congenital or traumatic injury involving either limb
* patients already on selenium medication
* patients participating in another clinical study related to lymphedema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2004-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of orally administered selenium compared to placebo in reducing arm lymphedema in patients treated with surgery (axiallary nodal dissection) and radiotherapy for breast cancer.

SECONDARY OUTCOMES:
To assess the toxicity of selenium.
To assess the association of selenium, quality of life and limb function.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Levin, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada